CLINICAL TRIAL: NCT00657904
Title: A Randomized Double-Blind Comparative Trial of Bicalutamide (Casodex™) Versus Placebo in Patients With Early Prostate Cancer.
Brief Title: Bicalutamide (Casodex™) Versus Placebo in Patients With Early Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D6876C00023; 7054IL/0023
Record Dates: First submitted 2008-04-07; First posted 2008-04-14 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Non-metastatic Prostate Cancer
Keywords: androgen antagonists; prostate neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Bicalutamide
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bicalutamide — 150mg daily
  Other Names: Casodex™
  Arms: 1
Drug: Placebo — once daily
  Arms: 2

SUMMARY:
The purpose of this trial is to study the effect - in terms of time to progression and overall survival - of 2 years of adjuvant bicalutamide 150mg monotherapy, versus placebo, in subjects with histologically or cytologically confirmed non-metastatic adenocarcinoma of the prostate gland.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer in the early stage of disease
* Prostate removed and/or radiation therapy to the prostate area

Exclusion Criteria:

* Previous systemic therapy for prostate cancer
* Previous history of another form of cancer (not prostate) within 5 years of study start.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3618 (Actual)
Dates: Start 1995-08; Primary Completion 2008-07 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Time to clinical progression | Throughout study period
Overall patient survival | Throughout study period

SECONDARY OUTCOMES:
Time to treatment failure | Throughout study period
Serum prostate-specific antigen | Initial study period up to 2006 amended protocol
Tolerability in terms of adverse events and laboratory parameters | Throughout study period

CONTACTS AND LOCATIONS:
Overall Officials: William See, Principal Investigator — Medical College of Wisconsin; David G. McLeod, Principal Investigator — Walter Reed Army Medical Center
Locations (85):
- United States (72):
  - Research Site, Birmingham, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Scottsdale, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Berkeley, California
  - Research Site, Laguna Woods, California
  - Research Site, Newport Beach, California
  - Research Site, San Diego, California
  - Research Site, San Francisco, California
  - Research Site, Santa Monica, California
  - Research Site, Thousand Oaks, California
  - Research Site, Torrance, California
  - Research Site, Van Nuys, California
  - Research Site, Denver, Colorado
  - Research Site, Middlebury, Connecticut
  - Research Site, New Haven, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Aventura, Florida
  - Research Site, Bay Pines, Florida
  - Research Site, Boca Raton, Florida
  - Research Site, Daytona Beach, Florida
  - Research Site, Fort Myers, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Miami, Florida
  - Research Site, Ocala, Florida
  - Research Site, Saint Augustine, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Fort Wayne, Indiana
  - Research Site, Greenwood, Indiana
  - Research Site, Iowa City, Iowa
  - Research Site, Kansas City, Kansas
  - Research Site, Louisville, Kentucky
  - Research Site, Shreveport, Louisiana
  - Research Site, Greenbelt, Maryland
  - Research Site, Rockville, Maryland
  - Research Site, Burlington, Massachusetts
  - Research Site, Newtown, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, Hattiesburg, Mississippi
  - Research Site, Jackson, Mississippi
  - Research Site, St Louis, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, Lebanon, New Hampshire
  - Research Site, Albany, New York
  - Research Site, Manhasset, New York
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Syracuse, New York
  - Research Site, The Bronx, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Lancaster, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Cordova, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Danville, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Virginia Beach, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Madison, Wisconsin
  - Research Site, Milwaukee, Wisconsin
  - Research Site, Cheyenne, Wyoming
- Canada (13):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Victoria, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Halifax, Nova Scotia
  - Research Site, Hamilton, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, London, Ontario
  - Research Site, North York, Ontario
  - Research Site, Oakville, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec

REFERENCES:
- [Derived] Iversen P, McLeod DG, See WA, Morris T, Armstrong J, Wirth MP; Casodex Early Prostate Cancer Trialists' Group. Antiandrogen monotherapy in patients with localized or locally advanced prostate cancer: final results from the bicalutamide Early Prostate Cancer programme at a median follow-up of 9.7 years. BJU Int. 2010 Apr;105(8):1074-81. doi: 10.1111/j.1464-410X.2010.09319.x. PMID 22129214